CLINICAL TRIAL: NCT03016377
Title: Administration of Autologous CAR-T Cells Targeting the CD19 Antigen and Containing the Inducible caspase9 Safety Switch in Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia
Brief Title: Administration of Autologous CAR-T CD19 Antigen With Inducible Safety Switch in Patients With Relapsed/Refractory ALL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Bellicum Pharmaceuticals (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1541-ATL
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia; Immune System Diseases; Immunoproliferative Disorders
Keywords: CAR T cells; CD19; Leukemia; T Lymphocytes; AP1903; Cytokine Release Syndrome; Rimiducid; ICANS; Immune effector cell mediated neurotoxicity syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Immune System Diseases; Immunoproliferative Disorders; Leukemia; Cytokine Release Syndrome | interventions — AP 1903 reagent; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iC9-CAR19 cells (Experimental): The 3+3 design in adult subjects and an independent study using 3+3 design in pediatric subjects. The starting dose of 5 x 10^5 transduced cells/kg will enroll 3 adult subjects in the initial cohort. If there are no dose limiting toxicities w/in 4 weeks of the cell infusion in these 3 subjects, then the next cohort will evaluate 1 x10^6 transduced cells/kg in adults. If there is toxicity in 1/3 patients in the initial cohort, the cohort will be expanded to enroll up to 6 adult patients. If the dose level 1 is determined to be above the tolerated cell dose, de-escalation would occur to dose level -1 where subjects would receive 1 x 10^5 transduced cells/kg. All subjects will receive a lymphodepleting regimen of fludarabine and cyclophosphamide before administration of iC9-CAR19 T cells.
  Interventions: Biological: iC9-CAR19 cells; Drug: Rimiducid; Drug: Cyclophosphamide; Drug: Fludarabine
- Expansion Cohort Second Administration of iC9-CAR19 cells (Experimental): After the recommended phase 2 dose (RP2D) of iC9-CAR19 T cells has been determined in adults, up to 18 additional adult subjects will be enrolled in an expansion cohort at the RP2D. In the expansion cohort, subjects will be offered a second infusion of iC9-CAR19 T cells based on B-cell recovery and minimal residual disease (MRD) status. All subjects will receive a lymphodepleting regimen of fludarabine and cyclophosphamide before second administration of iC9-CAR19 T cells.
  Subjects in the expansion cohort who experience ≥grade 2 CRS or ICANS, did not respond to the initial dose of the standard of care treatment will be enrolled in a sub-study of rimiducid.
  Interventions: Biological: iC9-CAR19 cells; Drug: Rimiducid; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: iC9-CAR19 cells — Three dose levels are being evaluated: dose level -1 (1 x 10^5), dose level 1 (5 x 10^5), and dose level 2 ( 1x 10^6)
  Other Names: CAR.CD19 T cells
Drug: Rimiducid — Subjects with CRS and ICAN will assign one of two dose levels (DL)s of rimiducid with the standard treatment: 0.05 mg/kg or 0.1 mg/kg for subjects with CRS and 0.01mg/kg or 0.1mg/kg for subjects with ICAN. Subjects will first be enrolled on DL 1 and then enrolled on DL 2, and 0.4mg/kg rimiducid will be given to subjects who did not respond to the initial dose.
  Other Names: AP1903
Drug: Cyclophosphamide — 900 mg/m^2 IV over 1 hour on day 4 of lymphodepleting chemotherapy.
  Other Names: Neosar
Drug: Fludarabine — 25 mg/m^2/day IV over 30 minutes administered for 3 consecutive days.
  Other Names: Fludara

SUMMARY:
The body has different ways of fighting infection and disease. No single way is effective at fighting cancer. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are proteins that protect the body from disease caused by bacteria or toxic substances. Antibodies work by binding those bacteria or substances, which stops them from growing and causing bad effects. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected. Both antibodies and T cells have been used to treat patients with cancers. They both have shown promise, but neither alone has been sufficient to cure most patients. This study combines both T cells and antibodies to try to create a more effective treatment. This investigational treatment is called autologous T lymphocyte chimeric antigen receptor cells targeted against the CD19 antigen (ATLCAR.CD19) administration.

In previous studies, it has been shown that a new gene can be put into T cells that will increase their ability to recognize and kill cancer cells. A gene is a unit of DNA. Genes make up the chemical structure carrying the genetic information that may determine human characteristics (i.e., eye color, height and sex). The new gene that is put in the T cells makes a piece of an antibody called anti-CD19. This antibody can flow through the blood and can find and stick to leukemia cells because these leukemia cells have a substance on their surface called CD19. Anti-CD19 antibodies have been used to treat people with leukemia but have not been strong enough to cure most patients. For this study, the anti-CD19 antibody has been changed so that instead of floating free in the blood a piece of it is now joined to the surface of the T cells. Only the part of the antibody that sticks to the leukemia cells is attached to the T cells instead of the entire antibody. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These CD19 chimeric (combination) receptor-activated T cells kill some of the tumor, but they do not last very long in the body and so their chances of fighting the cancer are unknown.

Preliminary results of giving ATLCAR.CD19 cells to leukemia patients have been encouraging; however, many subjects receiving this treatment have experienced unwanted side effects including neurotoxicity and/or cytokine release syndrome (also referred to as cytokine storm or an infusion reaction). Cytokines are small proteins that interreact as e signals to other cells and are the way cells talk to one another. During cytokine release syndrome, too many cytokines are released and too many cells in your body react to their release. Symptoms resulting from cytokine release syndrome vary from flu-like symptoms to more severe side effects such as cardiac arrest, multi-system organ failure or death. We predict that about 50% of patients on this study will experience mild to severe cytokine release syndrome.

To help reduce cytokine release syndrome symptoms in future patients, a safety switch has been added to the ATLCAR.CD19 cells that can cause the cells to become dormant or "go to sleep". The safety switch is called inducible caspase 9 or iC9. The modified ATLCAR.CD19 cells with the safety switch are referred to as iC9-CAR19 cells.

The purpose of this study is to determine whether receiving the iC9-CAR19 cells is safe and tolerable (there are not too many unwanted effects). Researchers has previously tested different doses of the iC9-CAR19. An effective dose that had the least number of unwanted side effects in patients was identified. It was planned to test this dose in more patients to learn more about its effect in the body. This type of research study is called a dose expansion study. It will allow the investigators to collect more information about the effect of this dose in treating of certain type of cancer.

DETAILED DESCRIPTION:
LCCC1541-ATL is a Phase I/Phase II dose finding trial to determine if chimeric antigen receptor T (CAR-T) cells targeting the CD19 antigen and containing the inducible caspase 9 safety switch can be safely administered to adult and pediatric subjects with relapsed or refractory CD19+ acute lymphoblastic leukemia (ALL).

OUTLINE

Cell Procurement

Peripheral blood, up to 300 mL total (in up to 3 collections) will be obtained from subjects for cell procurement. In subjects with inadequate lymphocyte count in the peripheral blood, a leukopheresis may be performed to isolate sufficient T cells. The parameters for apheresis will be up to 2 blood volumes.

Lymphodepleting Regimen

Subjects will receive a lymphodepleting regimen of fludarabine 25 mg/m2/day administered IV over 30 min for three consecutive days and a single IV dose of cyclophosphamide 900 mg/m2 administered over 1 hour on the fourth day. If iC9-CAR19 T cell infusion is delayed for >4 weeks, lymphodepletion may be repeated prior to iC9-CAR19 T cell infusion.

Administration of iC9-CAR19 T Cells

Post lymphodepletion, subjects who meet eligibility criteria for cellular therapy will receive iC9-CAR19 T cells within 2-14 days after completing the pre-conditioning chemotherapy regimen. We will administer iC9-CAR19 post lymphodepletion at dose levels specified. A phase I trial performed by Lee et al established that 1×106 CAR19+ T cells/kg was safe and associated with significant in vivo expansion and we anticipate similar results with iC9-CAR19+ T cells.

Second Cell Infusion Requirements:

Subjects will be offered a second infusion based on B-cell recovery and MRD status >4 weeks after the initial infusion if cells are available or if the subject has sufficient stored peripheral blood to manufacture additional iC9-CAR19 T cells.

Duration of Therapy

Therapy in LCCC1541-ATL involves 1 infusion of iC9-CAR19 cells. Treatment with one infusion will be administered unless:

* Subject decides to withdraw from study treatment, or
* General or specific changes in the subject's condition render the subject unacceptable for further treatment in the judgment of the investigator.

A second infusion with prior lymphodepletion will be given to subjects enrolled in the expansion cohort and to subjects enrolled in the dose escalation cohort once the RP2D is reached if they meet the eligibility requirements for lymphodepletion and infusion. Specifically, only subjects with the following characteristics will be offered a second infusion:

* B-cell recovery (defined as absolute CD19+ cell count >50/μL in the blood or bone marrow within 6 months of initial infusion AND/OR
* MRD positive (defined as ≥0.01% as assessed by multi-parameter flow cytometry) with CD19+ expression at any time after the initial infusion.
* *Note that subjects who receive dose level 1 in the dose escalation will receive the RP2D for their second infusion, if applicable.

Duration of Follow-up

Subjects will be followed for up to 15 years after the final iC9-CAR19 T-cell infusion for RCR evaluation or until death, whichever occurs first. Subjects removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

Subjects who receive new therapy (such as hematopoietic stem cell transplant) after a cell product administration will still be required to complete abbreviated follow up procedures.

ELIGIBILITY:
All clinical and laboratory data required for determining eligibility must be available in the subject's medical/research record which will serve as the source document. Subjects may be transfused with blood products to obtain a hemoglobin level > 7.0 g/dL and platelet count > 20,000 per μl.

Note: During the period after cell procurement and during iC9-CAR19 T-cell production, subjects are allowed to receive standard of care intervening therapy for ALL to manage their disease if the treating physician feels it is in the subject's best interest Common Inclusion Criteria for all subjects

* Written informed consent for procurement signed by the subject or the legal guardian of a pediatric subject and HIPAA authorization
* Age 3 to 17 years of age for pediatric subjects (weight must be ≥10 kg), ≥ 18 to 70 years of age for adults at the time of consent.
* Karnofsky score > 60%, if ≥16 years old, or Lansky performance score of greater than 60% if <16 years old .

Demonstrate adequate renal and hepatic function as defined below; all screening labs to be obtained within 72 hours prior:

System Laboratory Value Renal* Serum Creatinine (sCr) ≤ 1.5 × ULN) Hepatic: Total bilirubin (tBili) ≤ 1.5 × ULN, unless attributed to Gilbert's Syndrome Aspartate aminotransferase (AST) ≤ 3.0 × ULN Alanine aminotransferase (ALT) ≤ 3.0 × ULN

* Females of childbearing potential must have a negative serum pregnancy test within 72 hours prior to procurement. Note: Females are considered of childbearing potential unless they are premenarchal, surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Females and males of childbearing potential must be willing to abstain from heterosexual activity or to use two forms of effective methods of contraception from the time of informed consent until 3 months after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method. Female participants will inform their male partners that they must use the methods of birth control required by the protocol.
* Male subjects with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 3 months after the last dose of study therapy. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures.

Inclusion Criteria for Cell Procurement

* Relapsed or refractory precursor B cell ALL:

  * 2nd or greater bone marrow or central nervous system (CNS) relapse,
  * Any bone marrow or CNS relapse >100 days after allogeneic stem cell transplant, Primary refractory ALL defined as no complete response after 2 cycles of a standard of care chemotherapy regimen, or
  * For adult subjects: first bone marrow or CNS relapse with duration of first CR <1 year, or CR1 duration ≥1 year and refractory to ≥1 cycle of therapy for treatment of relapse
  * Subjects with isolated non-CNS extramedullary disease will be eligible as long as the time-of-remission criteria above for bone marrow and CNS relapses or primary refractory ALL are met and the biopsy for extramedullary disease confirms CD19 expression
  * For pediatric subjects: first bone marrow, CNS or isolated non-CNS extramedullary relapse refractory to more than 1 cycle of standard therapy for relapsed ALL
  * While active CNS3 leukemia will be excluded, subjects with concurrent CNS3 disease and bone marrow relapse who have responded to CNS-directed therapy prior to enrollment will be allowed to participate. Intrathecal chemotherapy will be allowed to continue between lymphodepleting chemotherapy and cell infusion.
  * Subjects with CNS2 disease and concurrent bone marrow relapse will be eligible. Intrathecal chemotherapy will be allowed to continue between lymphodepleting chemotherapy and cell infusion
  * Subjects who have previously achieved remission with no detectible measurable residual disease (MRD) by multi-parameter flow cytometry, and who have re- developed CD19+ MRD measured by multi-parameter flow cytometry will be eligible, provided that the duration of first MRD-negative CR was <1 year, MRD- negative CR1 duration ≥1 year and refractory to ≥1 cycle of therapy for treatment of MRD recurrence, or MRD reappearance occurs during second or subsequent CR.
  * Subjects who have persistent CD19+ MRD measured by multi-parameter flow cytometry after 3 cycles of initial chemotherapy, and have persistence of CD19+ MRD after one or more cycles of blinatumomab.
* Subjects with Ph+ ALL will be eligible if they have failed ≥ 2 ABL tyrosine kinase inhibitors, relapsed after allogeneic stem cell transplant or have CD19+ MRD. Subjects with the T315I ABL kinase point mutation will be eligible if they have failed ponatinib-containing therapy, regardless of the number of prior ABL tyrosine kinase inhibitors.
* CD19 positivity of lymphoblasts confirmed by flow cytometry or IHC per institutional standards.
* Life expectancy ≥ 12 weeks.
* Demonstrate adequate renal and hepatic function as defined below; all screening labs to be obtained within 72 hours prior to procurement.

  *For pediatric patients, adequate renal function is defined as below: Age Maximum Serum Creatinine (mg/dL) Both (Male, Female) 3 to <6 years ≤0.8 6 to <10 years ≤1 10 to <13 years ≤1.2 13 to <16 years (Male) ≤1.5 / Female ≤1.4 16 to <18 years (Male) ≤1.7 / Female ≤1.4
* Subjects currently receiving "maintenance" doses of chemotherapy are eligible and the need for intrathecal prophylaxis prior to procurement is left to the discretion of the investigator. Maintenance doses of systemic chemotherapy are defined as methotrexate ≤30 mg/m2/week, mercaptopurine ≤100 mg/m2/day and vincristine ≤ 2 mg/28 days. Maintenance therapy in patients with Ph+ leukemia may also contain tyrosine kinase inhibitors (TKIs) targeting BCR-ABL, at the discretion of the investigator. Corticosteroid- containing maintenance therapy is permitted only if corticosteroids are administered >14 days prior to procurement.

Exclusion Criteria for Cell Procurement

Subjects meeting any of the following criteria cannot be enrolled in this study:

* Subjects with relapsed fulminant CD19+ ALL that is rapidly progressing with circulating lymphoblasts that are rising in proportion to >50% of circulating white blood cells.
* Intrathecal chemotherapy will be allowed to continue between cell procurement and lymphodepleting chemotherapy.
* Pregnant or breastfeeding (Note: breast milk cannot be stored for future use if the milk is collected while the mother is being treated on study).
* Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
* Subjects must not have tumor in a location where enlargement could cause airway obstruction.
* Subjects may not have an oxygen requirement as defined by pulse oximetry of <90% on room air.
* Subjects must not have left ventricular ejection fraction of <40% (shortening fraction <27% for pediatric subjects) as measured by echocardiogram or MUGA.
* Patients with the following systemic viral infections will be excluded: active HIV, HBV, HCV. Only subjects meeting the criteria as so described will be infused. Note: To meet eligibility subjects are required to be negative for HIV antibody or HIV viral load, negative for Hepatitis B surface antigen, or negative for HCV antibody or HCV viral load
* Patients who are on treatment for other active uncontrolled infections (not referenced above) with resolution of signs/symptoms are not excluded. Non-influenza, non-RSV, isolated upper respiratory infections are not excluded. Other active uncontrolled infections will be excluded.
* Prior to procurement current use of systemic corticosteroids at doses ≥10 mg/day prednisone or its equivalent; those receiving <10 mg/day may be enrolled at discretion of investigator. (Note: Corticosteroid use with doses at the discretion of the treating physician are allowed after procurement up to the beginning of lymphodepletion. Corticosteroid use is contraindicated following iC9-CAR19 infusion unless medically necessary e.g., to treat CRS).
* Physiologic replacement with hydrocortisone is allowed at doses 6-12 mg/m2/day, or equivalent.
* Received anti-CD19 antibody-based therapy or cytotoxic chemotherapy not described as maintenance therapy (within 2 weeks of procurement per section).

Inclusion Criteria for Lymphodepletion:

* Relapsed or refractory precursor B cell ALL, confirmed by presence of blasts in the blood or bone marrow (≥5%) or in any extramedullary site. Subjects who have previously achieved remission with no detectible measurable residual disease (MRD) by multi- parameter flow cytometry, and who have re-developed CD19+ MRD measured by multi- parameter flow cytometry are eligible, provided that the duration of first MRD-negative CR was <1 year, MRD-negative CR1 duration ≥1 year and refractory to ≥1 cycle of therapy for treatment of MRD recurrence/relapse, or MRD-recurrence in second or subsequent morphologic CR. Additionally, subjects who have persistent CD19+ MRD measured by multi-parameter flow cytometry after 3 cycles of initial chemotherapy, and have persistence of CD19+ MRD after one or more cycles of blinatumomab are eligible to participate. Because CNS leukemia is not curable with conventional therapies, subjects who met inclusion criterion for CNS leukemia at the time of procurement will be eligible for lymphodepletion even if intrathecal or systemic chemotherapy has rendered their cerebrospinal fluid free of lymphoblasts prior to lymphodepletion.
* Life expectancy ≥ 12 weeks.
* Subjects who have received prior therapy with murine antibodies must have documentation of absence of human anti-mouse antibodies (HAMA) prior to lymphodepletion on this study.

Demonstrate adequate renal and hepatic function as defined below; all screening labs to be obtained within 72 hours prior to lymphodepletion.

* For pediatric patients, adequate renal function is defined as below:

Age Maximum Serum Creatinine (mg/dL) Both Male/Female 3 to <6 years ≤0.8 6 to <10 years ≤1 10 to <13 years ≤1.2 13 to <16 years (Male) ≤1.5/ (Female) ≤1.4 16 to <18 years (Male) ≤1.7/(Female) ≤1.4

* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures.
* For subjects who receive chemotherapy between cell procurement and lymphodepletion, washout periods as described in exclusion criteria sections 4.4.5 to 4.4.11 between chemotherapy and the beginning of lymphodepletion will be required.
* Subjects must have autologous transduced activated T cells that meet the Certificate of Analysis (CofA) acceptance criteria.

Exclusion Criteria for Lymphodepletion

Subjects meeting any of the following criteria cannot be enrolled in this study:

* Pregnant or breastfeeding (Note: breast milk cannot be stored for future use if the milk is collected while the mother is being treated on study).
* Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
* Subjects must not have tumor in a location where enlargement could cause airway obstruction.
* Subjects may not have an oxygen requirement as defined by pulse oximetry of <90% on room air.
* Treatment with any investigational drug within 14 days (i.e., two weeks) prior to lymphodepletion or has received any tumor vaccines within the previous five weeks prior to lymphodepletion.
* Subject has received pegylated-asparaginase ≤3 weeks prior to lymphodepletion.
* Radiotherapy to a non-CNS site completed <1 week prior to lymphodepletion, or CNS directed radiation completed <7 weeks prior to lymphodepletion.
* Subject is receiving following drugs <1 week prior to lymphodepletion: salvage chemotherapy (e.g. clofarabine, cytosine arabinoside > 100 mg/m2, anthracyclines, cyclophosphamide, methotrexate ≥ 25 mg/m2)..
* Any systemic drug used for GVHD must be stopped >3 weeks prior to lymphodepletion (e.g. calcineurin inhibitors, methotrexate or other chemotherapy drugs, mycophenolyate, rapamycin, thalidomide, or immunosuppressive antibodies such as anti-CD20 (rituximab), anti-TNF, anti-IL6 or anti-IL6R, systemic steroids).
* The following drugs must be stopped prior to the beginning of lymphodepleting chemotherapy: tyrosine kinase inhibitors, hydroxyurea, vincristine, 6-mercaptopurine, 6- thioguanine, methotrexate <25 mg/m2, cytosine arabinoside <100 mg/m2/day, and asparaginase (non-pegylated). These drugs should not be administered concomitantly or following lymphodepleting chemotherapy .
* CNS prophylaxis or treatment of CNS leukemia with intrathecal methotrexate, cytarabine and/or hydrocortisone treatment must be stopped prior to lymphodepleting chemotherapy.
* Patients with the following systemic viral infections will be excluded: active HIV, HTLV, HBV, HCV. Note: To meet eligibility subjects are required to be negative for HIV antibody or HIV viral load, negative for Hepatitis B surface antigen, or negative for HCV antibody or HCV viral load.
* Patients who are on treatment for other active uncontrolled infections (not referenced above) with resolution of signs/symptoms are not excluded. Non-influenza, non-RSV, isolated upper respiratory infections are not excluded. Other active uncontrolled infections will be excluded.
* Use of systemic corticosteroids at doses ≥10 mg/day prednisone or its equivalent; those receiving <10 mg/day may be enrolled at discretion of investigator. (Note: Corticosteroid use with doses at the discretion of the treating physician are allowed after procurement up to the beginning of lymphodepletion.).

Physiologic replacement with hydrocortisone is allowed at 6-12 mg/m2/day, or equivalent.

Inclusion Criteria- iC9-CAR19 Cell Infusion

* Subjects must fulfill all of the following inclusion criteria to participate in this study:
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures.

Exclusion Criteria- iC9-CAR19 Cell Infusion

* Subjects meeting any of the following criteria cannot be enrolled in this study:
* Corticosteroid use is contraindicated following iC9-CAR19 infusion unless medically necessary (e.g., to treat CRS).
* Severe systemic uncontrolled disease or toxicities that develop after lymphodepletion may prompt exclusion from cell infusion at the discretion of the investigator.
* Received any donor lymphocyte infusions (DLI) ≤6 weeks prior to iC9-CAR19 T cell product administration.
* Received any T cell lytic or toxic antibody (e.g. alemtuzumab) ≤8 weeks prior to iC9- CAR19 T cell product administration (residual lytic levels may destroy the infused iC9- CAR19 T cells and/or prevent their in vivo expansion).

Inclusion Criteria Prior to Lymphodepletion for the Second Infusion

* Life expectancy ≥ 12 weeks.
* Documentation of absence of human anti-mouse antibodies (HAMA). Demonstrate adequate renal and hepatic function as defined below; all screening labs to be obtained within 72 hours prior to lymphodepletion.

Subject meets at least one of the following criteria:

* B-cell recovery (defined as absolute CD19+ cell count of >50/μL in the blood or bone marrow CD19+ B cells ≥0.5% of marrow aspirate cells by flow cytometry) within 6 months of initial infusion. Subjects who meet this criteria within 6 months of initial infusion may be started on lymphodepletion at a date later than 6 months from initial infusion.
* MRD positive (defined as ≥0.01% as assessed by multi-parameter flow cytometry) with CD19+ expression at any time after initial infusion.
* At least 4 weeks have passed since the initial iC9-CAR19 T cell infusion.
* Subjects have resolved/recovered symptoms from CRS and/or ICANS that developed after prior iC9-CAR19 T cell infusion.
* Subjects must have autologous transduced activated T cells that meet the Certificate of Analysis (CofA) acceptance criteria. The subject must have sufficient available cells or have sufficient stored peripheral blood to manufacture additional iC9-CAR19 T cells.

Exclusion Criteria for Lymphodepletion for the Second Infusion

Subjects meeting any of the following criteria cannot receive a second infusion as part of this study:

* Pregnant or breastfeeding (Note: breast milk cannot be stored for future use if the milk is collected while the mother is being treated on study).
* Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
* Subjects must not have tumor in a location where enlargement could cause airway obstruction.
* Subjects may not have an oxygen requirement as defined by pulse oximetry of <90% on room air.
* Patients who are on treatment an active uncontrolled infections with resolution of signs/symptoms are not excluded. Non-influenza, non-RSV, isolated upper respiratory infections are not excluded. Other active uncontrolled infections will be excluded.
* Use of systemic corticosteroids at doses ≥10 mg/day prednisone or its equivalent; those receiving <10 mg/day may be enrolled at discretion of investigator. (Note: Corticosteroid use with doses at the discretion of the treating physician are allowed after procurement up to the beginning of lymphodepletion.).

Physiologic replacement with hydrocortisone is allowed at 6-12 mg/m2/day, or equivalent.

Inclusion Criteria- Second iC9-CAR19 Cell Infusion

Subjects must fulfill all of the following inclusion criteria to receive a second iC9- CAR19 cell infusion on this study:

Exclusion Criteria- Second iC9-CAR19 Cell Infusion

Subjects meeting any of the following criteria cannot receive a second iC9-CAR19 cell infusion on this study:

* Corticosteroid use is contraindicated following iC9-CAR19 infusion unless medically necessary (e.g., to treat CRS).
* Severe systemic uncontrolled disease or toxicities that develop after lymphodepletion may prompt exclusion from cell infusion at the discretion of the investigator

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-03-22 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2037-09-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of iC9-CAR19 T cells | 4 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (AEs) (CTCAE, version 5.0), a descriptive terminology which can be utilized for AE reporting. A grading (severity) scale is provided for each AE term/symptom: Grade 1 (Mild; asymptomatic); Grade 2 (Moderate; minimal, local or noninvasive intervention indicated); Grade 3 (Severe or medically significant but not immediately life-threatening; hospitalization indicated; disabling); Grade 4 (Life-threatening consequences; urgent intervention indicated); Grade 5 (Death related to AE). Immune effector cell-associated neurotoxicity syndrome (ICANS) symptoms will be graded according to the criteria outlined in the protocol on a scale from 1 (mild) to 4 (critical). Cytokine release syndrome (CRS) will be graded according to criteria outlined in the protocol on a scale from 1 (mild) to grade 5 (death).

SECONDARY OUTCOMES:
Incidence of dose limiting toxicity to identify recommended phase 2 dose (RP2D) | 4 weeks
  The recommended phase 2 dose of iC9-CAR19 cells in adult and pediatric subjects will be determined maximum dose at which no more than one out of six patients experiences a dose limiting toxicity (DLT). A DLT is defined according to protocol criteria using the NCI CTCAE, ICANS, and CRS criteria. In general, a DLT is any grade 3 or higher event that is at least possibly related to iC9-CAR19 T cells.
Changes in persistence of iC9-CAR19 T cells in vivo | 15 years
  Persistence of iC9-CAR19 T cells in vivo will be determined by quantitative polymerase chain reaction (PCR) and flow cytometry in samples of peripheral blood.
Overall Response Rate (ORR) | 15 years
  ORR (Complete Response/Complete Response with incomplete recovery of counts) to first iC9-CAR19 T cell therapy will be determined using National Comprehensive Cancer Network Response Criteria (NCCN) for acute lymphoblastic leukemia. Assessment of minimal residual disease will be included as criterion of response (ie, the percentage of subjects who achieve CRm [defined as minimal residual disease negative complete response] by either flow cytometry or PCR analysis will be determined)
Overall survival after infusion of iC9-CAR19 T cells | 15 years
  Overall survival will be measured from the date of administration of first iC9-CAR19 T cells to the date of death.
Event-free survival rate | 15 years
  Event free survival rate applies to all subjects and will be measured from the date of administration of first iC9-CAR19 T cells to the date of signs and symptoms of treatment failure or relapse from complete response or complete response with incomplete recovery of counts, or death from any cause; subjects not known to have any of these events are censored on the date they were last examined.
Relapse-free survival rate | 15 years
  Relapse-free survival rate will apply only to subjects achieving complete response or complete response with incomplete recovery of counts and measured from the date of achievement of a remission until the date of relapse or death from any cause; subjects not known to have relapsed or died at last follow-up are censored on the date they were last examined.
Incidence of patient reported symptoms in adult patients using selected symptoms from the NCI PRO-CTCAE | 15 years
  The NCI Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) is a patient-reported outcome measurement system developed to characterize the frequency, severity and interference of 78 symptomatic treatment toxicities.
Changes in patient reported physical functions in adult patients | 15 years
  Patient reported physical functions in adult patients will be assessed per the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Score derived from the PROMIS Physical Function Short Form 20a v1.0. PROMIS is a set of person-centered measures, developed by the US Department of Health and Human Services, that evaluates and monitors physical, mental, and social health on a five point Likert scale with higher score indicating better functioning.
Changes in patient reported health-related quality of life in adult patients | 15 years
  Patient reported health-related quality of life will be assessed using the PROMIS (Patient-Reported Outcomes Measurement Information System) Global Health Score derived from the PROMIS Global Health Short Form v1.0-1.1. PROMIS is a set of person-centered measures, developed by the US Department of Health and Human Services, that evaluates and monitors physical, mental, and social health health on a five point Likert scale with higher score indicating better functioning.
Number of participants with adverse events as a measure of safety and tolerability of a second infusion of iC9-CAR19 T cells | 4 weeks
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (AEs) (CTCAE, version 5.0), a descriptive terminology which can be utilized for AE reporting. A grading (severity) scale is provided for each AE term/symptom: Grade 1 (Mild; asymptomatic); Grade 2 (Moderate; minimal, local or noninvasive intervention indicated); Grade 3 (Severe or medically significant but not immediately life-threatening; hospitalization indicated; disabling); Grade 4 (Life-threatening consequences; urgent intervention indicated); Grade 5 (Death related to AE). Immune effector cell-associated neurotoxicity syndrome (ICANS) symptoms will be graded according to the criteria outlined in the protocol on a scale from 1 (mild) to 4 (critical). Cytokine release syndrome (CRS) will be graded according to criteria outlined in the protocol on a scale from 1 (mild) to grade 5 (death).
Rate of measurable residual disease (MRD) clearance in subjects who receive iC9-CAR19 T cells for MRD persistence or MRD-only relapse | 8 weeks
  Rate of MRD clearance will be defined as the proportion of subjects who enter MRD-negative complete response (CRm) who are treated with one or two infusions of iC9 CAR19 T cells at the time of being in complete response (CR) or Complete Response with incomplete recovery of counts (CRi), but not CRm.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie S Grover, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://unclineberger.org/patientcare/clinical-trials/clinical-trials